CLINICAL TRIAL: NCT01401634
Title: Oral Hydration for Mild to Moderate Hyperglycemia in the Emergency Department
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sanjay Arora MD, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10-00223
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Hyperglycemia
Keywords: Hyperglycemia Hydration
MeSH Terms: conditions — Hyperglycemia | interventions — Water

ARMS (2):
- Intravenous Fluids (Other): Intravenous fluids for patients with hyperglycemia is part of the standard protocol in our department
  Interventions: Other: Intravenous normal saline
- Oral Fluids (Experimental)
  Interventions: Other: Oral water

INTERVENTIONS:
Other: Oral water — 2 Liters of water given orally
  Arms: Oral Fluids
Other: Intravenous normal saline — 2 Liters Intravenous normal saline
  Arms: Intravenous Fluids

SUMMARY:
Diabetes and high blood sugar are extremely common among patients presenting to US Emergency Departments. Intravenous fluids with or without insulin are often used to treat these patients. However, simple, low-cost interventions, such oral hydration have not been studied in this context. Oral rehydration may be better than no therapy at all, which is often what these patients receive in the first few hours when presenting to busy, overcrowded Emergency Department (ED) with long wait times, or in resource-poor environments such as developing countries. The investigators propose a study to see if oral hydration for adult patients presenting to the ED with high blood sugar i.e. finger-stick (FS) values between 250 and 500 mg/dL can help lower blood sugar at the same rate as intravenous fluids. Half the patients will be given intravenous fluids per our department protocol, while the other half of the patients will be given 2 liters of water to drink over a 1-hour period. Both groups will have their blood sugar measured every 30 mins for 2 hours. The investigators will analyze the data to determine if there is a statistically significant difference in blood sugar between the two groups within 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Any patient, above the age of 18 years old, presenting to Emergency Department triage with a fingerstick glucose between 250 and 500 mg/dL

Exclusion Criteria:

* Patients with evidence of DKA (hyperglycemia with ketonuria and abnormal pH or bicarbonate on venous blood gas), HHS, or other critical illnesses requiring immediate medical attention (as determined by ED triage nurses),
* end-stage renal disease requiring dialysis through an arterio-venous shunt or fistula,
* abnormal mental status (GCS < 15),
* unstable vital signs including pulse > 100, SBP < 100, respiratory rate>20, (or any combination of vital signs not meeting these cutoffs but deemed worrisome by the triage nurse) or unable to tolerate oral intake/actively vomiting.
* Patients who receive IV fluids prior to or during the study period.
* Patients unable to communicate in English or Spanish.
* Jail patients will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in Blood Sugar | 2 hours
  Patients will have their blood sugar checked every 30 minutes for 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States